CLINICAL TRIAL: NCT00198770
Title: Does Substitution of Meat Products With White Button Mushrooms Have Potential for Weight Reduction? Studies of the Level of Short and Intermediate-term Caloric Compensation, Satiety, and Dietary Satisfaction Among Lean and Obese Men and Women.
Brief Title: Dietary Compensation With Substitution of Meat Products With White Button Mushrooms.
Acronym: Mush 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Mushroom Council (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: MC2004-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Crossover design - 1 arm (Experimental): Meat week followed by mushroom week, counterbalanced order
  Interventions: Dietary Supplement: dietary substitution to assess level of caloric compensation

INTERVENTIONS:
Dietary Supplement: dietary substitution to assess level of caloric compensation — Mushrooms substituted for meat in dishes

SUMMARY:
Unfortunately, current methods of achieving weight control are disappointing. There is also a great deal of public confusion over what constitutes an appropriate diet for weight control; there is a paucity of carefully performed, randomized, controlled clinical treatment trials to evaluate the varying opinions. Mushrooms are not widely appreciated as the nutritious, low calorie, low fat food (and potential meat substitute) that they are. Mushrooms may be a new "diet food," especially as a substitute for higher calorie and fat staples like meat.

This study examines whether there is compensation for the potential calorie and fat savings of substituting mushrooms for meat in dishes over a 4-day period.

DETAILED DESCRIPTION:
1. Development of suitable mushroom-meat substitutions. In this phase, guided by information gathered from test subjects (see 2. below) we will devise and internally taste-test test meals that entail mushroom substitutions that result in potential energy savings of at least 125 kcal per meal.
2. Study the palatability, consumer acceptance, and satiating properties of each mushroom-substituted meal using a panel of obese and normal weight men, women, seniors, and teenagers.
3. Test in a controlled fashion the percent compensation over a 4-day period for the calorie and fat deficit that results when these mushroom-substituted meals are consumed compared with unsubstituted meals among obese and normal weight adults.

In this phase, the following two hypotheses will be tested:

Hyp 1. Use of white button mushrooms as a substitute for meat at a single meal will result in significant reduction in total daily energy intake during the same 24 h period.

Hyp 2. The amount of calories and fat grams compensated for will be significantly less than 100% when the substitution of mushrooms for meat is continued on a one-meal daily basis for a period of 4 days.

Summary of experimental design: Controlled intervention study, crossover design with each subject serving as his or her own control. Subjects: n=40 healthy men and women, aged 18-65, stratified by BMI Intervention: 11-day feeding study divided into two, 4-day intervention periods (Mondays through Thursdays), separated by a 3-day washout period (Friday through Sunday); subjects fed a standard lunch meal on site, and precise food records gathered for any meals or snacks taken off-site. One of the two 4-day intervention periods will include one meal per day that substitutes one of the 7 mushroom meals devised in phases 1 and 2 in place of meat meals, while the other 4-day intervention period will be the same except for not having any substituted meals. The order of the interventions will be randomized to eliminate order effects. Satiety measures will be obtained as in experiment #3, as well as measures of diet satisfaction. Weight will be measured.

ELIGIBILITY:
Inclusion Criteria:

ages 18-65 (for phase 3), Body Mass Index between 18-45; not using appetite-affecting medications unless on established and stable dose; not using weight loss drugs; willing and able to comply with the protocol requirements; willing and able to give informed consent.

Exclusion Criteria:

Those participants that: have a strong dislike of the foods that may be involved; have a mold allergy/food allergy; have chronic, uncontrolled health problems (not including obesity and diabetes); have bulimia, laxative abuse, substance abuse, alcohol intake > 10 drinks per week, or have an uncontrolled psychiatric disorder (major depression, bipolar disorder, etc as determined at screening); are breast-feeding or pregnant at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-03; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Total energy intake- by meal, by day separately for days 1-4, and by total intervention period (mushroom substituted vs. not) | 2 wks
Percent calorie and fat-gram compensation- again by meal, day, and period. | 2 wks

SECONDARY OUTCOMES:
Satiety (VASs)- by meal, day, and period. | 2 wks
All outcomes will be analyzed for the total study population, and separately by gender and weight class. | 2 wks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Cheskin LJ, Davis LM, Lipsky LM, Mitola AH, Lycan T, Mitchell V, Mickle B, Adkins E. Lack of energy compensation over 4 days when white button mushrooms are substituted for beef. Appetite. 2008 Jul;51(1):50-7. doi: 10.1016/j.appet.2007.11.007. Epub 2007 Dec 3. PMID 18221822